CLINICAL TRIAL: NCT01328782
Title: The Post-Operative Pain Management of Pediatric Supracondylar Elbow Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-1190
Record Dates: First submitted 2010-09-22; First posted 2011-04-05 (Estimated); Results first posted 2012-06-13 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2012-06

CONDITIONS: Elbow Fracture
Keywords: elbow fracture; supracondylar elbow fracture; elbow; fracture; pain management; pediatric
MeSH Terms: conditions — Elbow Fractures; Fractures, Bone; Agnosia | interventions — Oxycodone; Acetaminophen; oxycodone-acetaminophen; Bupivacaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- The group receiving oral pain medicine (Active Comparator): This group will receive Oxycodone with Acetaminophen orally
  Interventions: Drug: Oxycodone with Acetaminophen
- The group receiving bupivacaine and oral pain medicine (Active Comparator): This group will receive an intra-articular shot during surgery and will then be sent to the recovery room to receive pain medication as needed.
  Interventions: Drug: Bupivacaine 0.25%
- The group receiving ropivacaine and oral pain medicine (Active Comparator): This group will receive an intra-articular shot of ropivacaine during surgery and will be sent to the recovery room to receive pain medicine as needed.
  Interventions: Drug: Ropivacaine 0.20%

INTERVENTIONS:
Drug: Oxycodone with Acetaminophen — 0.1- 0.15 mg/kg (oxycodone) every 4-6 hours as needed. Pills: 325 mg acetaminophen: 5 mg oxycodone per tablet. Liquid: 325 mg acetaminophen:5 mg oxycodone per 5 mL.
  Other Names: Percocet
  Arms: The group receiving oral pain medicine
Drug: Bupivacaine 0.25% — * Up to 4 ml at 0.25 % given to .. In toxic doses can lead to irregular heart beat, patients aged 4-7 (dose will be irregular heart rate and cardiac arrest. (This no greater than 0.71 mg/kg)
  * Up to 5 ml at 0.25 % by volume solution will be given to patients aged 8-12 (dose will be no greater than 0.63 mg/kg)
  * All doses given will be significantly less then maximum allowable dose of 2.5- 3.0 mg/kg
  Other Names: Marcaine
  Arms: The group receiving bupivacaine and oral pain medicine
Drug: Ropivacaine 0.20% — * Up to 4 ml at 0.20 % given to patients aged 4-7 (dose will be no greater than 0.57 mg/kg)
  * Up to 5 ml at 0.20 % by volume solution will be given to patients aged 8-1(dose will be no greater than 0.50 mg/kg)
  * All doses given will be significantly less then maximum allowable dose of 2.5- 3.0 mg/kg
  Other Names: Naropin
  Arms: The group receiving ropivacaine and oral pain medicine

SUMMARY:
The goal of this study is to compare different ways of treating pain after surgery. This research study involves subjects who have a supracondylar elbow fracture and need surgery. This type of fracture occurs when the humerus (upper arm bone) is broken just above the elbow. Like any other surgery, you can expect that you will feel pain in the hours or days after the operation. Currently, despite the common occurrence of this surgery, there is not a standard way to treat and or prevent any of the pain afterwards.

At this hospital, oral (take by mouth) pain medicine is commonly used to treat pain after this surgery.

In this study, pain will be treated in one of the following ways:

1. with oral pain medication
2. with oral pain medicine and an intraarticular shot (a shot into the elbow joint) of bupivacaine (a "numbing" drug) or
3. with oral pain medicine and an intraarticular shot of ropivacaine (another "numbing" drug). The shots will be given during surgery. Your participation will help us find out which of these three pain control methods works the best.

The correct dosages of all drugs will be safely prescribed by the doctor on an individual basis and all drugs will be used under the careful watch of your attending physician. All the drugs used this study are approved by the FDA for use in adults but they are not specifically approved for use in children. However, nearly 7 out of every 10 drugs approved for adults are not specifically approved by the FDA for use in children. All drugs used in this study will be used in a way that is considered to be safe and reasonable by the Children's Hospital.

DETAILED DESCRIPTION:
Purpose: In recent years, despite the lack of consistent evidence, the use of intraarticular (into the joint)injections during ambulatory, orthopaedic surgery has become a popular strategy for reducing post-operative pain. In this randomized, single center, prospective study the investigators will evaluate the analgesic effectiveness of intraarticular injections of local anesthesia during the closed reduction and percutaneous pinning (CRPP) of supracondylar type elbow fractures (SCEFx) in children. In order to determine the efficacy of intraarticular injections, perceived post-operative pain will be compared among the three study groups receiving either a 0.25 % intraarticular injection of bupivacaine (Group 1 ), a 0.20% intraarticular injection of ropivacaine (Group 2) or no intraarticular injection (Control). All groups will receive the same post-operative oral pain medication of oxycodone (0.1 to 0.15 mg/kg) with acetaminophen.

Primary Aim(s) : Compare the primary and secondary pain outcomes variables in each of the three study groups.

* The primary pain outcome variables are defined as the following:

  * Self-reported pain within 30-60 min. of arrival to the recovery room
  * Self-reported pain at two hours post-operative
* The secondary pain outcome variables are defined as the following:

  * Parent perception of post-operative pain (scores of modified version of Foster and Varni's Total Quality of Pain Management Survey (TQPM) given in the first two hours after surgery)
  * Time t o first administration of oral pain medication
  * Total dose and frequency of oral pain medication taken during first 72 hours post-operative
  * Dose (per kg) of local anesthetic received intra-operatively
  * Total dosage of all intra-operative analgesics (in morphine equivalents)
  * Pre-operative The Faces Pain Scale-Revised (FSP-R) score

Hypotheses for Primary Aims:

* There will not be a significant difference in any of the pain outcome variables amongst Groups 1 and 2.
* There will be a statistically significant difference in each of the pain outcome variables when comparing; Group 1 and Control as well as Group 2 and Control.

Secondary Aim I: Evaluate the overall effect gender, ethnicity, age, American Society of Anesthesiologists (ASA) classification, fracture type and anesthesia time have on the pain outcome variables in this study population:

Hypotheses for Secondary Aim I: The investigators expect that age, gender, ASA classification, fracture type and anesthesia time will have a significant effect of on the primary and secondary pain outcome variables in this study population as a whole.

* Participants aged 4-7 will be associated with more pain than participants aged 8-12 (increased selfreported pain scores, increased parent TQPM scores, decreased time to first administration of oral pain medication, increased total dosage of oral pain medication taken during first 72 hours post-operative, increased frequency of oral pain medication taken during first 72 hours post-operative).
* Females will be associated with more pain than males (increased self-reported pain scores, increased parent TQPM scores, decreased time to first administration of oral pain medication, increased total dosage of oral pain medication taken during first 72 hours post-operative, increased frequency of oral pain medication taken during first 72 hours post-operative ) .
* An ASA classification of III will be associated with more pain than a classification of I or II (increased self-reported pain scores, increased parent TQPM scores, decreased time to first administration of oral pain medication, increased total dosage of oral pain medication taken during first 72 hours post-operative, increased frequency of oral pain medication taken during first 72 hours post-operative),
* A type III fracture type will be associated with more pain than a type I or II (increased selfreported pain scores, increased parent TQPM scores, decreased time to first administration of oral pain medication, increased total dosage of oral pain medication taken during first 72 hours post-operative, increased frequency of oral pain medication taken during first 72 hours post-operative).
* An increase in anesthesia time will be associated with more pain . (increased self-reported pain scores, increased parent TQPM scores, decreased time to first administration of oral pain medication, increased total dosage of oral pain medication taken during first 72 hours post-operative, increased frequency of oral pain medication taken during first 72 hours post-operative).

Secondary Aim II: Evaluate the overall effect that gender, ethnicity, age, ASA classification (I, II or III),fracture type and anesthesia time have on the pain outcome variables in each of the study groups (Compare 1, 2 and Control to study population as a whole).

Hypotheses for Secondary Aim II: The investigators anticipate that there will be no group difference in the effects that age, gender, ASA classification, fracture type or anesthesia time have on the primary and secondary pain outcome variables.

Secondary Aim III: Compare Group 1 and Group 2 for a potential dose dependent relationship between reported pain outcome variables and total dose of intraarticular injection.

Hypotheses for Secondary Aim III: In both groups, the investigators anticipate there will be a non-significant association between an increased dose of local anesthetic and decreased post-operative FSP-R scores. There will not be any difference in the significance of this dose dependent relationship between Group I and Group 2.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I, II or III
* Patients 4-12 years old requiring general anesthesia for closed reduction and percutaneous pinning (CRPP) of supracondylar type elbow fractures (SCEFx).
* Patients able to understand and report their pain with the Faces Pain Scale Revised

Exclusion Criteria:

* Medical contraindications to analgesic therapy.
* Known allergy or sensitivity to analgesic agent.
* Clinical evidence of skin inflammation precluding the 'clean' area at the site of injection.
* Patients lacking the cognitive understanding to report their pain with the FSP-R (unable to complete seriation task).
* Patients necessitating open reduction due to inability to obtain an acceptable closed reduction.
* Comorbid diagnosis of other traumatic injury that causes any local and or global pain.
* Patients presenting to ER with neurovascular injury or compartment syndrome due to fracture.
* For patients in either of the two intervention arms, if after three attempts, the intraarticular injection is not successful, the patient will be dropped from the study.
* Patients admitted for complications directly related to the surgery will be dropped from analysis. Any such event will be immediately reported to COMIRB with in five business days. However, patients admitted due to a late afternoon/evening surgery and patients admitted for standard observational purposes unrelated to surgical complications, will not be dropped from the study.
* Known drug allergy to oxycodone and or acetaminophen.
* Children 4-7 years old weighing less than 14 kg (Weight exclusion criteria is based on a 4 year old female that is below the fifth percentile for weight, per the Center for Disease Control Growth Charts).
* Children 8-12 years old weighing less than 20 kg (Weight exclusion criteria based on an 8 year old female that is below the fifth percentile for weight, per the Center for Disease Control Growth Charts).

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Narcotic Group: This group will receive Oxycodone with Acetaminophen orally
- Bupivacaine Group: This group will receive an intra-articular shot during surgery and will then be sent to the recovery room to receive pain medication as needed.
- Ropivacaine Group: This group will receive an intra-articular shot of ropivacaine during surgery and will be sent to the recovery room to receive pain medicine as needed.
Period: Overall Study
Arm/Group | Oral Narcotic Group | Bupivacaine Group | Ropivacaine Group
Started | 43 | 42 | 39
Completed | 43 | 42 | 39
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Narcotic Group | Bupivacaine Group | Ropivacaine Group | Total
Number analyzed (Participants) | 43 | 42 | 39 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 43 | 42 | 39 | 124
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.92 (1.99) | 6.86 (1.74) | 6.73 (2.21) | 6.85 (1.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 18 | 54
  Male | 25 | 24 | 21 | 70
Region of Enrollment [Number; unit: participants]
  United States | 43 | 42 | 39 | 124

OUTCOME MEASURES:

1. Primary Outcome: The Faces Pain Scale-Revised (FSP-R) Scores (Scored 0-10).
Description: The Faces Pain Scale Revised is a dimensionless 10 point likert scale used to assess self-reported pain intensity on a scale from 0 (no pain) to 10 (most pain you can imagine). Greater pain scores are indicative of more severe pain.
Time Frame: Will be obtained 30 - 60 minutes after arrival to the recovery room
Population: Based on the number of participants that self-reported their pain score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Oral Narcotic Group | Bupivacaine Group | Ropivacaine Group
Number analyzed (Participants) | 37 | 41 | 35
Scores on a scale | 4.14 (3.45) | 2.73 (3.28) | 3.66 (3.58)
Statistical Analysis 1: Comparison: Oral Narcotic Group vs Bupivacaine Group; Test type: Superiority or Other; p = 0.074, ANOVA; Mean Difference (Net) = 1.40, 95% CI [1.40 to 2.94]
Statistical Analysis 2: Comparison: Bupivacaine Group vs Ropivacaine Group; Test type: Superiority or Other; p = 0.556, ANOVA; Mean Difference (Final Values) = 0.556, 95% CI [-1.12 to 2.08]
Statistical Analysis 3: Comparison: Oral Narcotic Group vs Ropivacaine Group; Test type: Superiority or Other; p = 0.244, ANOVA; Mean Difference (Final Values) = 0.93, 95% CI [-0.64 to 2.49]

2. Secondary Outcome: Total Quality Pain Management Survey (TQPM) Scores for Questions # 16: Child's Current Level of Pain, Question # 17: Child's Worst Level of Pain When Moving Around After Surgery and Question # 18: Child's Worst Level of Pain While Resting
Description: Total quality pain management survey is validated survey used to assess parents' perceptions of their child's pain. Pain is assessed on a dimensionless 10 pt likert scale from 0 (no pain) to 10 (severe pain). Greater pain scores are indicative or more severe pain.
Time Frame: Will be obtained from parent(s) 120 minutes after arrival to the recovery room
Population: Based on number of participants and their parents/legal guardians that completed the survey.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Oral Narcotic Group | Bupivacaine Group | Ropivacaine Group
Number analyzed (Participants) | 38 | 37 | 37
Scores on a scale | 4.58 (3.40) | 2.73 (2.58) | 4.32 (3.22)
Statistical Analysis 1: Comparison: Oral Narcotic Group vs Bupivacaine Group; Test type: Superiority or Other; p = 0.014, ANOVA; Mean Difference (Final Values) = 1.81, 95% CI 2-sided [0.38 to 3.25]
Statistical Analysis 2: Comparison: Oral Narcotic Group vs Ropivacaine Group; Test type: Superiority or Other; p = 0.832, ANOVA; Mean Difference (Net) = 0.16, 95% CI [-1.30 to 1.61]
Statistical Analysis 3: Comparison: Bupivacaine Group vs Ropivacaine Group; Test type: Superiority or Other; p = 0.027, ANOVA; Mean Difference (Final Values) = 1.66, 95% CI [0.20 to 3.12]

3. Secondary Outcome: Time (in Minutes) to First Narcotic Administration
Time Frame: first 72 hours after surgery close time
Population: All subjects were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Oral Narcotic Group | Bupivacaine Group | Ropivacaine Group
Number analyzed (Participants) | 43 | 42 | 39
Minutes | 30 [20.5 to 53.5] | 50.5 [30.5 to 115.3] | 34 [21.5 to 56.5]
Statistical Analysis 1: Comparison: Oral Narcotic Group vs Bupivacaine Group; Test type: Superiority or Other; p = 0.005, Log Rank
Statistical Analysis 2: Comparison: Oral Narcotic Group vs Ropivacaine Group; Test type: Superiority or Other; p = 0.3767, Log Rank
Statistical Analysis 3: Comparison: Bupivacaine Group vs Ropivacaine Group; Test type: Superiority or Other; p = 0.039, Log Rank

4. Secondary Outcome: Total Dosage in Morphine Equivalents (mg/kg) of All Analgesics Received in Prior to Discharge
Time Frame: Analgesic data collected during first four hours following the end of surgery (surgery close)
Population: All subjects were included in the analysis.
Measure: Mean (Standard Deviation); unit: Morphine (po) equivalents [mg*kg-1]
Arm/Group | Oral Narcotic Group | Bupivacaine Group | Ropivacaine Group
Number analyzed (Participants) | 43 | 42 | 39
Morphine (po) equivalents [mg*kg-1] | 0.09 (0.09) | 0.05 (0.05) | 0.08 (0.09)
Statistical Analysis 1: Comparison: Oral Narcotic Group vs Bupivacaine Group; Test type: Superiority or Other; p = 0.008, ANOVA; Mean Difference (Final Values) = 0.042, 95% CI [0.008 to 0.076]
Statistical Analysis 2: Comparison: Bupivacaine Group vs Ropivacaine Group; Test type: Superiority or Other; p = 0.078, ANOVA; Mean Difference (Final Values) = 0.031, 95% CI [-0.004 to 0.066]
Statistical Analysis 3: Comparison: Oral Narcotic Group vs Ropivacaine Group; Test type: Superiority or Other; p = 0.5321, ANOVA; Mean Difference (Final Values) = 0.011, 95% CI [-0.024 to 0.045]

5. Secondary Outcome: Need for IV Morphine of Fentanyl
Description: Indicates that number of subjects that were in severe pain and thus required IV morphine and/or fentanyl.
Time Frame: First 120 minutes after the end of surgery (surgery close time)
Population: All subjects were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Oral Narcotic Group | Bupivacaine Group | Ropivacaine Group
Number analyzed (Participants) | 43 | 42 | 39
participants | 19 | 4 | 15
Statistical Analysis 1: Comparison: Oral Narcotic Group vs Bupivacaine Group; Test type: Superiority or Other; p = 0.004, Chi-squared
Statistical Analysis 2: Comparison: Bupivacaine Group vs Ropivacaine Group; Test type: Superiority or Other; p = 0.004, Chi-squared
Statistical Analysis 3: Comparison: Oral Narcotic Group vs Ropivacaine Group; Test type: Superiority or Other; p = 0.499, Chi-squared

ADVERSE EVENTS:
Arm/Group | Oral Narcotic Group | Bupivacaine Group | Ropivacaine Group
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/39
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No